CLINICAL TRIAL: NCT03279406
Title: REgistry on Real-Life EXperience With Left Atrial Appendage Occlusion for Patients With Atrial Fibrillation in France
Brief Title: REgistry on Real-Life EXperience With Left Atrial Appendage Occlusion
Acronym: RELEXAO
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Principal Investigator, Laurent Fauchier, Professor of Cardiology, University Hospital, Tours
Other Study IDs: Cardio Tours RELEXAO
Record Dates: First submitted 2017-09-06; First posted 2017-09-12 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Stroke; Thrombus; Left atrial appendage; Bleeding
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Thrombosis; Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Percutaneous Left Atrial Appendage Occlusion — Percutaneous left atrial appendage occlusion in routine care for patients with atrial fibrillation

SUMMARY:
The objective of this observational non-randomized multicenter study is to compile real-world clinical characteristics and outcomes data for patients treated with LAA (left atrial appendage) closure systems in a daily clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are eligible for a LAA occlusion device and treated with a commercially available device according to international and local guidelines and per physician discretion.

Exclusion Criteria:

* None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated with percutaneous Left Atrial Appendage Occlusion among those referred to one of the French centers involved in this database
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | From date of inclusion until the date of first documented event, whichever came first, assessed up to 60 months
  Death, Ischemic stroke, Transient ischemic attack, Major hemorrhage, Thrombus on device

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Fauchier, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Tours

REFERENCES:
- [Derived] Fauchier L, Cinaud A, Brigadeau F, Lepillier A, Pierre B, Abbey S, Fatemi M, Franceschi F, Guedeney P, Jacon P, Paziaud O, Venier S, Deharo JC, Gras D, Klug D, Mansourati J, Montalescot G, Piot O, Defaye P. Device-Related Thrombosis After Percutaneous Left Atrial Appendage Occlusion for Atrial Fibrillation. J Am Coll Cardiol. 2018 Apr 10;71(14):1528-1536. doi: 10.1016/j.jacc.2018.01.076. PMID 29622159